CLINICAL TRIAL: NCT03848546
Title: Vezel-UP:Stimulating Fiber Intake Via Personalized Dietary Advice
Brief Title: Stimulating Fiber Intake Via Personalized Dietary Advice
Acronym: Vezel-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Netherlands: Ministry of Health, Welfare and Sports (Other Government); Dutch Association for Gastrointestinal diseases (MLDS) (Unknown); Bolletje (Unknown); Sensus (Industry); Sonneveld (Unknown); Kellogg Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NL67998.028.18
Record Dates: First submitted 2019-01-22; First posted 2019-02-20 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Dietary Habits; Dietary Fiber; Personalized Advice; Microbiota
Keywords: fiber intake; personalized dietary advice; stool pattern; perceived wellbeing
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Two groups: one receives general advice (control), the other personalized advice (intervention). Subjects are followed over time.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PDA (Experimental): Intervention group: receives the personalized dietary advice
  Interventions: Behavioral: PDA
- Control (Active Comparator): Receives the general advice (two flyers containing information about fiber intake)
  Interventions: Other: Control (no intervention)

INTERVENTIONS:
Behavioral: PDA — Subjects receive personal dietary fiber advice to increase their fiber intake. This advice will be provided using an online web-portal, where subjects can choose high-fiber alternatives that closely match their own intake. The aim is to "swap" product for low in fiber for a high fiber alternative (such as white bread, whole wheat bread).
  Arms: PDA
Other: Control (no intervention) — No intervention
  Arms: Control

SUMMARY:
Dietary fibers are linked to improved health and prevention of diseases such as obesity, stroke, hypertension, diabetes and colorectal cancer. Moreover, fibers play a crucial role in improving and maintaining gut health, by increasing stool weight,stool frequency and improvement of stool consistency. Currently, very few adults meet the recommendation of 30 (females) or 40 (males) grams per day. Personalized dietary advice may be the solution to increase dietary fiber intake in large populations.

The objective is to investigate if a personalized dietary advice is more effective in increasing dietary fiber intake in the Dutch population than the general advice that is currently provided by the Netherlands Nutrition center and the Dutch Digestive Foundation (MLDS).Second objective is to assess the effect of increased fiber intake on stool pattern, perceived well-being and consumer behavior parameters and the role of psychological factors in the effectiveness of personalized dietary advice on dietary fiber intake.

Study design: A 4.5-month (6 weeks intervention + follow-up after 3 months) single-blind randomized controlled trial with two groups: the intervention group, which receives personalized dietary advice (PDA), and the control group, which only receives the general dietary advice. Primary study parameters/outcome of the study: Primary endpoint is dietary fiber intake, which will be assessed using an Food Frequency Questionnaire and 24hr recalls.

Fecal microbiota composition and metabolite levels will be used as an objective marker for fiber intake. Secondary study parameters/outcome of the study (if applicable):

Secondary parameters include stool pattern, well-being, hunger, satiety and body weight. Furthermore, psychological measurements will give insight into why the PDA was (not) effective.

DETAILED DESCRIPTION:
This study is performed in healthy adults, older than 18 years, with no gastro-intestinal complaints. The intervention group receives personalized dietary advice (PDA) based on their current food pattern, preferences and selfregulation capacity. The PDA aims to compute high-fiber alternatives for products that subjects currently use and that are close to their current eating behavior, to help increase dietary fiber intake. This PDA will be provided using an online webportal. The control group only receives a general dietary advice, e.g. (a) flyer(s) containing information on fibers from the Netherlands Nutrition Center and the MLDS. The intervention group will also receive this general advice next to the PDA.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Apparently healthy: no gastrointestinal complaints, no food allergies and no medication that can influence the outcome of the study (see exclusion criteria).
* Relatively low fiber intake: which is assessed by a short fiber intake screening questionnaire (score ranging from

  1 to 22). Females with a score ≤13 and males with a score ≤15 will be included in the study.
* Living in the surroundings of Wageningen (max. 50 km).
* In possession of a mobile phone with android ≥4.4 or iOS system ≥9 to use apps.
* Signed informed consent.

Exclusion Criteria:

* Any digestive tract disorder that is expected to interfere with the study outcomes, such as chronic constipation or diarrhea, Crohn's Disease, Ulcerative Colitis, Irritable Bowel Syndrome, Coeliac disease.
* Diagnosis of Diabetes Mellitus, since the change in carbohydrate intake may interfere with medication usage.
* Currently following a strict diet and unwilling or unable to change; for example a gluten free diet or a "crash diet" using meal substitutes.
* Use of medication that can interfere with the study outcomes, including laxatives, diuretics, antidepressants, codeine, antibiotics or fiber supplements
* Female subjects: currently pregnant or breastfeeding, or intending to become pregnant during the study, as this can affect stool patterns and well-being.
* Simultaneously participating in another study.
* Unwilling or unable to fulfill the study criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-09-14 (Actual); Study Completion 2019-09-14 (Actual)

PRIMARY OUTCOMES:
Change in dietary fiber intake | Before study, after 6 weeks intervention, and 3 months follow-up
  Will be measured using the Food Frequency Questionnaire, and 24hr recalls to compute grams of fiber.
change in Short Chain Fatty acid level | Before study, at 3 weeks and at 6 weeks
  of a fecal sample
change in Microbiota composition | Before study, at 3 weeks and at 6 weeks
  of a fecal sample

SECONDARY OUTCOMES:
Stool pattern | Daily during 6-week intervention
  Bristol stool chart en stool frequency
Perceived wellbeing | Daily during 6-week intervention
  Using validated questions
Hunger and Satiety | Daily during 6-week intervention
  Using validated questions
Body weight | study start, and after 6 weeks
  Subjects weigh themselves (morning, fasted)
Psychological questionnaires | Before and after the 6-week intervention, and at 3-months follow-up
  Validated questionnaire will be used to assess motives, barriers, knowledge, intentions, self-efficacy, self-regulation and knowledge

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University, Division of Human Nutrition, Wageningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rijnaarts I, de Roos N, Zoetendal EG, de Wit N, Witteman BJM. Development and validation of the FiberScreen: A short questionnaire to screen fibre intake in adults. J Hum Nutr Diet. 2021 Dec;34(6):969-980. doi: 10.1111/jhn.12941. Epub 2021 Aug 29. PMID 34378249
- [Derived] Rijnaarts I, de Roos NM, Wang T, Zoetendal EG, Top J, Timmer M, Bouwman EP, Hogenelst K, Witteman B, de Wit N. Increasing dietary fibre intake in healthy adults using personalised dietary advice compared with general advice: a single-blind randomised controlled trial. Public Health Nutr. 2021 Apr;24(5):1117-1128. doi: 10.1017/S1368980020002980. Epub 2020 Sep 18. PMID 32943128